CLINICAL TRIAL: NCT05490875
Title: A Pilot Study of Carotid Ultrasound to Identify Head and Neck Cancer Survivors With High Cardiovascular Risk After Radiation Therapy
Brief Title: Carotid Ultrasound to Identify Head and Neck Cancer Survivors With High Cardiovascular Risk After Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00087922; WFBCCC 98322 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer; Carotid Artery Stenosis; Cardiovascular Complication
MeSH Terms: conditions — Head and Neck Neoplasms; Carotid Stenosis | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood (total 16 mL) will be obtained from patients who opt to provide these samples. Plasma and peripheral blood mononuclear cells (PBMC) will be banked for the following planned correlative analyses, pending further funding. Upon collection, these samples will be collected (see Correlative Blood Specimen Collection Form), transported to and processed/stored by the NCORP Biorepository for future analysis. If funding is not obtained for correlative studies by the closure of this study, samples will be retained indefinitely for future study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid Ultrasound Group: Head and neck cancer survivors treated with radiotherapy, at least 2 years since end of radiotherapy with no evidence of disease will receive a carotid ultrasound to measure carotid velocities and intima-media thickness of the carotid arteries.
  Interventions: Procedure: Carotid ultrasound; Other: Blood draw; Other: Survey

INTERVENTIONS:
Procedure: Carotid ultrasound — Carotid ultrasound will be done to both sides of the neck to look at the carotid arteries.
Other: Blood draw — This optional blood draw could occur anytime from the time of enrollment on the study until 90 days after the research ultrasound.
Other: Survey — Participants will complete a 15-minute survey about how acceptable participants find the ultrasound procedure, whether participants would be open to it in the future if a doctor thought it was necessary, whether participants would be open to getting treatment for artery problems, and how participants feel about their own risk of stroke.

SUMMARY:
The purpose of this research study is to understand how radiation therapy may affect blood vessels in the neck called the carotid arteries. Investigators want to look at narrowing of the artery or thickening of the walls of the arteries.

DETAILED DESCRIPTION:
Primary Objective: To determine the proportion of patients with clinically significant carotid artery stenosis (≥50% stenosis) in head and neck cancer survivors treated with head and neck radiotherapy.

Secondary Objectives:

* To measure the intima-media thickness (IMT) of the carotid arteries in head and neck cancer survivors treated with head and neck radiotherapy.
* To determine the proportion of patients with carotid intima-media thickness of at least 0.9 mm in head and neck cancer survivors treated with head and neck radiotherapy.
* To determine the proportion of patients with carotid plaque of maximum thickness 2 mm or greater in head and neck cancer survivors treated with head and neck radiotherapy.
* To determine the proportion of patients identified as having a high risk of cardiovascular events (relative risk 1.50 or greater) based on intima-media thickness measurements in head and neck cancer survivors treated with head and neck radiotherapy.
* To describe the risk of significant carotid artery stenosis based on various clinical factors in head and neck cancer survivors treated with head and neck radiotherapy.
* To determine the feasibility of carotid ultrasound in head and neck cancer survivors treated with head and neck radiotherapy.
* To obtain preliminary data on the acceptability of carotid ultrasound among head and neck cancer survivors treated with head and neck radiotherapy.
* To obtain preliminary data on barriers to potential carotid ultrasound screening in head and neck cancer survivors treated with head and neck radiotherapy.
* To obtain preliminary data on stroke risk perception among head and neck cancer survivors treated with radiotherapy in head and neck cancer survivors treated with head and neck radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* History of head and neck cancer treated with radiotherapy. Radiotherapy target volume(s) must have included at least one region of the neck to a total dose of at least 45 gray (Gy).
* At least 2 years since completion of radiotherapy with no evidence of disease at the time of last clinical follow-up.
* Eligible by Screening Questionnaire.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Personal history of any of the following: Carotid artery stenosis on either side of the neck, stroke (CVA) or transient ischemic attack (TIA), carotid endarterectomy, carotid stent placement.
* Prior carotid artery ultrasound examination between completion of radiotherapy and registration.
* Most recent radiotherapy treatment was for any recurrence of a prior head and neck cancer and/or treatment for a subsequent head and neck cancer after diagnosis and treatment of an initial head and neck cancer.
* Any history of re-irradiation to the head and neck region. Re-irradiation is defined as a subsequent individual course of radiotherapy where the target overlaps a region of the head/neck that was previously targeted by the initial course of radiotherapy.
* ECOG Performance Status of 2 or greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be screened through the radiation oncology clinic and by review of the electronic medical record for visits with head and neck radiation therapy providers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with 50% Stenosis Identified | At study completion, up to 1 approximately year
  This will be defined as having a peak systolic flow velocity of 150 cm/s or higher on Doppler ultrasonography will be estimated and reported along with an exact 95% confidence interval.

SECONDARY OUTCOMES:
Change in Intima-Media Thickness (IMT) | At time of ultrasound, up to approximately 1 year
  Mean, median, standard deviation and interquartile range will be used to describe IMT as a continuous variable at three separate angles (anterior, lateral and posterior). IMT will be measured in millimeters at 3 separate angles (anterior, lateral, and posterior) at the level of the distal common carotid artery, carotid bulb at the flow divider, and the proximal internal carotid artery.
Number of Participants with Carotid Intima-Media Thickness (IMT) Increase | At time of ultrasound, up to approximately 1 year
  Participants with at least one carotid IMT measurements of 0.9 mm or greater based on IMT measurements will be each be estimated and reported along with an exact 95% confidence interval.
Number of Participants with Carotid Plaque Thickness Increase | At time of ultrasound, up to approximately 1 year
  Participants with carotid plaque of maximum thickness 2 mm or greater and with high risk of cardiovascular events (relative risk 1.50 or greater) based on IMT measurements will be each be estimated and reported along with an exact 95% confidence interval.
Number of Participants Identified at High Risk of Cardiovascular Events | At time of ultrasound, up to approximately 1 year
  Participants identified as clinically significant (relative risk 1.50 or greater) may be estimated and reported along with an exact 95% confidence interval within subgroups defined by clinical characteristics.
Number of Participants with Clinically Significant Carotid Artery Stenosis (Greater than or Equal to 50%) Based on Potential Risk Factors | At time of ultrasound, up to approximately 1 year
  Associations between continuous clinical characteristics and clinically significant carotid artery stenosis will be evaluated using t-tests or Wilcoxon rank-sum tests. Potential risk factors used to evaluate will be gender; age; systolic blood pressure at time of ultrasound; history of cigarette smoking; history of prior cardiovascular disease; history of atrial fibrillation; left ventricular hypertrophy on echocardiogram; use of anti-hypertensive medication; radiation dose to the exposed carotid artery
Number of Participants Enrolled that Receive Study Intervention - Feasibility | At time of enrollment, up to approximately 1 year
  The study will be considered feasible if 60% of responding participants enroll and receive carotid ultrasound. If less than 40% of responding participants enroll and receive the study carotid ultrasound, investigators will re-evaluate methods for subsequent study. This will be be reported with an exact 95% confidence interval.
Acceptability of Intervention Measure Instrument (Likert scale). | At study completion, up to approximately 1 year
  Descriptive statistics will be used to characterize acceptability of carotid ultrasound. Scoring scale is a Likert scale (completely disagree to completely agree) with completely agree being scored as a more positive response to the intervention and treatment options.
Barriers Survey instrument (Likert scale) | At study completion, up to approximately 1 year
  Descriptive statistics will be used to characterize barriers to getting a carotid ultrasound. Scoring scale is a Likert scale (completely disagree to completely agree) with completely agree being scored as a more positive response to the intervention and/or treatment options.
Assessment of Risk Perception Instrument (Likert scale) | At study completion, up to approximately 1 year
  Descriptive statistics will be used to characterize stroke risk perception. Scoring scale is a Likert scale (completely disagree to completely agree) with completely agree being scored as a more positive response to the intervention and/or treatment options.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hughes, MD, Principal Investigator — Wake Forest Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hughes RT, Snavely AC, Dressler EV, Tegeler CH, Nightingale CL, Furdui CM, Soto Pantoja DR, Register TC, Weaver KE, Lesser GJ. Carotid ultrasound to identify head and neck cancer survivors with high cardiovascular risk after radiation therapy: rationale and design of a prospective, cross-sectional pilot study. Future Oncol. 2024;20(31):2331-2341. doi: 10.1080/14796694.2024.2386927. Epub 2024 Sep 4. PMID 39230469